CLINICAL TRIAL: NCT05199610
Title: An Open-Label, Single-Dose, Parallel-Group Study of the Pharmacokinetics and Safety of EQ143 in Participants With Severe Hepatic Impairment and in Matched Healthy Adults
Brief Title: An Open-Label, Single-Dose, Parallel-Group Study of the Pharmacokinetics and Safety of EQ143
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EQRx International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EQ143-102
Record Dates: First submitted 2021-11-05; First posted 2022-01-20 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Severe Hepatic Impairment
MeSH Terms: interventions — aumolertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Aumolertinib (Experimental): single dose oral 55mg of aumolertinib
  Interventions: Drug: aumolertinib

INTERVENTIONS:
Drug: aumolertinib — A single dose of 55-mg EQ143 tablet will be administered in the morning on Day 1, and participants will remain for 5 days (4 nights) in the study center for collection of blood samples and safety monitoring. Participants will attend outpatient follow-up visits on Days 5, 6, 8, and 9 for additional blood sampling and safety assessments.
  Other Names: HS-10296

SUMMARY:
Participants aged 18 to 75 years with severe hepatic impairment (Child-Pugh class C) who meet the full study eligibility criteria will be enrolled into the study. For each participant with severe hepatic impairment, a corresponding healthy participant will be enrolled who matches with regard to age, sex, and BMI. A single dose of 55-mg EQ143 tablet will be administered in the morning on Day 1, and participants will remain for 5 days (4 nights) in the study center for collection of blood samples and safety monitoring. Participants will attend outpatient follow-up visits on Days 5, 6, 8, and 9 for additional blood sampling and safety assessments. The study will measure and describe the concentrations of EQ143 and its metabolite (HAS-719) in plasma over the course of 9 days (including calculation of PK parameters), the degree of EQ143 and metabolite HAS-719 (and other metabolites, if applicable) binding to proteins in plasma, and the safety of administering a single dose of EQ143 in severely hepatically impaired and matched healthy participants

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

Main Criteria for Inclusion: All Participants

1. Must be willing to participate in the study and sign the informed consent form (ICF).
2. Must be willing and able to complete all study-specific procedures and visits.
3. Is 18 to 75 years of age, inclusive, at Screening.
4. Is able to take and swallow oral medication.
5. BMI of 18.0 to 42.0 kg/m2
6. High probability for compliance with and completion of the study, in the opinion of the Investigator.
7. Must meet all of the applicable requirements for pregnancy and contraception, as follows:

   1. If female:

      * Is a female participant of childbearing potential who:

        * Has a negative serum pregnancy test result within 48 hours before Day -1;
        * Is not breastfeeding;
        * Agrees to use highly effective contraceptive measures during heterosexual intercourse throughout the study and for 12 weeks following EQ143 administration; AND
        * Agrees not to donate ova for the same time period; OR
      * Is a participant of non-childbearing potential, as confirmed by meeting both of the following criteria:

        * Has a negative serum or urine pregnancy test result within 48 hours before Day -1; AND is confirmed by the Investigator to be medically postmenopausal per one or more of the following parameters:

          * Age, in addition to any of the other parameters listed here;
          * Menses status (absence of menses for ≥ 1 year); or

            * Surgical status (prior hysterectomy, bilateral salpingectomy, or bilateral oophorectomy), with participant providing documentation of the surgical sterilization procedure (by operative report or ultrasound scan) prior to EQ143 administration; or
            * Follicle-stimulating hormone (FSH) level.
   2. If male:

      * Agrees to use a highly effective method of contraception (eg, male condom in addition to hormonal contraception) during heterosexual intercourse throughout the study and for 12 weeks following EQ143 administration; AND
      * Agrees to refrain from donating sperm for the same time period. Note: For all study participants, contraceptive use must be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

   Main Criteria for Inclusion: Hepatically Impaired Participants
8. Severe hepatic impairment (Child-Pugh class C according to the Child-Pugh classification).

   Notes:
   * Severe hepatic impairment is confirmed and documented based on at least one of the following: medical history, physical examination, computed axial tomography scan, magnetic resonance imaging and/or liver biopsy.
   * Screening laboratory test results for serum bilirubin; serum albumin; either activated partial thromboplastin time (aPTT) or prothrombin time (PT) (at site discretion); and stage of hepatic encephalopathy (with or without ascites) are consistent with Child-Pugh class C.
   * Hepatic impairment etiology should be one of the following: chronic alcoholism; chronic viral hepatitis; nonalcoholic steatohepatitis; autoimmune hepatitis; Wilson disease; alpha-1 antitrypsin deficiency; glycogen storage diseases; galactosemia; or cryptogenic.
9. If participant has concurrent stable medical condition(s) in addition to hepatic impairment-eg, diabetes without renal complications-the Investigator, Medical Monitor, and Sponsor Clinical Pharmacologist collectively agree that the condition(s) will not introduce an additional risk factor for the participant or interfere with the participant's ability to meet the study requirements.
10. If participant is taking medication(s) necessary for the management of their hepatic disease, and/or of concomitant stable medical conditions the medication regimen has been stable for at least 7 days before EQ143 administration and the Medical Monitor and Sponsor Clinical Pharmacologist agree that the medication is not expected to interfere with the PK of EQ143.

    Main Criteria for Inclusion: Healthy Matched Participants
11. Normal renal function, defined as calculated creatinine clearance ≥ 60 mL/min (as estimated by Cockroft-Gault equation).
12. Normal hepatic function, defined as total bilirubin ≤ 1.2 mg/dL and not meeting any Child-Pugh classification criteria
13. Healthy, as determined by the Investigator on the basis of medical history; physical examination; clinical laboratory test results; vital sign measurements; and 12-lead electrocardiogram (ECG).
14. Matched to the hepatically impaired participants in sex, age (± 10 years), and BMI (± 20% of BMI at Screening).

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

Main Criteria for Exclusion: All Medical History

1. Family history of QT prolongation, syncope, seizure, or unexplained cardiac-related death.
2. Presence or history of any disorder that may prevent the successful completion of the study.
3. Current or recent (within 3 months of Day 1 of the study) gastrointestinal disease that could impact the absorption of EQ143.
4. History of drug abuse within 1 year before Day 1 of the study
5. Is a regular smoker (ie, smokes more than 5 cigarettes per day or more than 10 packets per year), and is not willing to refrain from smoking from 48 hours before EQ143 administration through the final study visit.

   Allergies and Adverse Drug Reactions
6. History of any clinically important drug allergy or adverse drug reaction. Physical and Laboratory Findings
7. Plasma potassium and/or magnesium values outside the normal range.

   • Note: At the discretion of the Investigator, these tests may be repeated to confirm a result that is outside the normal range; repeat test results must be within normal limits to confirm participant eligibility.
8. An automatic ECG absolute QT interval with Fridericia's correction (QTcF) reading at Screening of > 480 ms (males) or > 500 ms (females).
9. Has evidence of active bacterial, fungal, or viral infection (including human immunodeficiency virus [HIV] or SARS-CoV-2, as detailed below) which would preclude safe enrollment as assessed by the treating Investigator.

   * Note regarding HIV: Participants with positive serologic finding and detectable HIV are excluded; however, participants with undetectable HIV and a viral load of 0 are not excluded if meeting all other eligibility criteria.
   * Note regarding SARS-CoV-2: The study SARS-CoV-2 requirements are determined by institutional standards (and local/country regulations, as applicable).

     * At Investigator discretion, any participant who tests positive and/or is symptomatic for SARS-CoV-2 during Screening may either be excluded from the study or delay enrollment until active infection has been excluded per institutional standards.
     * During the study, any SARS-CoV-2 testing is to be performed as clinically indicated for the individual participant. The Investigator must document the results of all tests performed. Any confirmed infection is to be recorded as an AE or, in the event that clinical manifestation warrants such, recorded and handled as an SAE as detailed.
10. Positive finding on urine drug screen (eg, amphetamines, barbiturates, benzodiazepines, cocaine, opiates), except a) cannabinoids or b) substances that are not prohibited per protocol and are legally prescribed to the participant, and have therefore been documented as concomitant medications (with additional considerations as noted below).

    • Note: Any participant who is taking any prescribed substance that triggers a positive urine drug screen result must have potential drug abuse ruled out by the Investigator. Additionally, any such participant must be confirmed by the Investigator to meet all other study eligibility criteria to rule out any potential excluded comorbidities associated with the prescribed substance.

    Prohibited Treatments
11. Consumption of alcoholic beverages from 24 hours before Day 1 of the study through the final study visit.
12. Consumption of grapefruit or grapefruit-containing products from 72 hours before Day 1 of the study through the final study visit.
13. Donation of blood within 30 days before Day 1 of the study.
14. Involvement in another investigational study of any type within 30 days before EQ143 administration

    Main Criteria for Exclusion: Hepatically Impaired Participants Medical History
15. Evidence of uncontrolled and clinically significant disease other than impaired hepatic function (eg, cardiovascular, gastrointestinal, cerebrovascular, respiratory, or renal disease, or any other comorbidity that, in the judgment of the Investigator, precludes participation in the study).
16. Has received, or is currently waiting for, an organ transplant.
17. Recent history or presence of any disorder that may interfere with the absorption, distribution, metabolism, or excretion of EQ143 (except those conditions associated with the hepatic disease) that may place the participant at risk during participation in the study, as assessed by the treating Investigator.
18. Presence of surgically created or transjugular intrahepatic portal systemic shunt.

    Physical and Laboratory Findings
19. Evidence of severe hepatorenal syndrome, as shown by calculated creatinine clearance < 40 mL/min (Cockroft-Gault equation).
20. Unstable liver disease, as shown by any of these factors/parameters:

    * Spontaneous bacterial peritonitis within 3 months before Day 1 of the study
    * Variceal bleeding within 1 month before Day 1 of the study
    * Severe hyponatremia (sodium level < 125 mmol/L)
    * Current evidence of hepatocellular cancer
    * Acute hepatic disease caused by an infection or drug toxicity
    * Severe encephalopathy (Grade 3-4 [Child-Pugh classification) unless at the time of Screening, it is controlled according to local standard of care (including ongoing treatment with lactulose)
    * Presence of severe ascites or severe edema that precludes participation in the study, as judged by the Investigator
    * Hemoglobin level ≤ 9.0 g/dL
    * Platelet count < 30 × 109/L for Child-Pugh class C participants
    * Total bilirubin level > 9 mg/dL
    * Relative increase of aPTT or PT by > 50% within the 2 weeks before EQ143 administration
    * Positive serologic findings for hepatitis B surface antigen (HBsAg) and/or hepatitis C virus (HCV) antibodies
    * Note: Test outcomes that are reactive to HCV antibody will be followed by an HCV ribonucleic acid (RNA) test (polymerase chain reaction [PCR]). Participants whose follow-up HCV RNA test (PCR) is reactive will be excluded.

    Prohibited Treatments
21. Prescription and over-the-counter (OTC) medication that is not taken according to a stable regimen for 7 days before EQ143 administration.
22. Use of any treatment known to be a strong CYP3A4 inhibitor or inducer within approximately 30 days or 5 half-lives, whichever is longer, before Day 1, with the exception of grapefruit or grapefruit-containing products (which are prohibited within 72 hours before Day 1 of the study, as noted above in Exclusion Criterion #12).
23. Use of any treatment known to be a sensitive CYP3A4 substrate within approximately 4 days (or 5 half-lives, whichever is longer) before and 4 days (or 5 half-lives, whichever is longer) after EQ143 administration.
24. Concomitant use of medications known to prolong the QTc interval.
25. Medications that alter gastric pH (eg, proton-pump inhibitors) within 3 days before and 2 days after EQ143 administration.

    Main Criteria for Exclusion: Healthy Matched Participants Medical History
26. Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.
27. Any surgical or medical condition that may interfere with the absorption, distribution, metabolism, or excretion of EQ143.
28. Acute disease state (eg, nausea, vomiting, fever, or diarrhea) within 7 days before Day 1 of the study.
29. . History of alcoholism within 1 year before Day 1 of the study, or consumption of more than 50 g of ethanol per day (12.5 cL glass of 10° [10%] wine = 12 g; 4 cL glass of aperitif; 42° [42%] whiskey = 17 g; 25 cL glass of 3° [3%] beer = 7.5 g; 25 cL glass of 6° [6%] beer = 15 g).

    Physical and Laboratory Findings
30. Any clinically significant findings on physical examination, vital sign measurements, 12-lead ECGs, or clinical laboratory test results.
31. Positive serologic findings for HBsAg and/or HCV antibodies.

    • Note: Test outcomes that are reactive to HCV antibody will be followed by an HCV RNA test (PCR). Participants whose follow-up HCV RNA test (PCR) is reactive will be excluded.

    Prohibited Treatments
32. Use of any prescription drug within 30 days or 5 half-lives, whichever is longer, before EQ143 administration, except hormone replacement therapy in postmenopausal female participants or treatments permitted in consultation with the Medical Monitor.
33. Use of any OTC drugs, including herbal supplements, within 14 days before Day 1 of the study, except for the occasional use of acetaminophen (paracetamol) and vitamins (≤ 100% of the recommended daily allowance).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) Parameter: Cmax of EQ143 | Predose and 1, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 168, and 192 hours post dose
  Cmax is defined as the maximum observed concentration of drug
PK Parameter: AUC0-t of EQ143 | Predose and 1, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 168, and 192 hours post dose
  AUC0-t is defined as the area under the concentration versus time curve from time zero to the last quantifiable concentration
PK Parameter: AUCinf of EQ143 | Predose and 1, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 168, and 192 hours post dose
  AUCinf is defined as the area under the concentration versus time curve extrapolated to infinite time
PK Parameter: CL/F of EQ143 | Predose and 1, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 168, and 192 hours post dose
  CL/F is defined as apparent clearance
PK Parameter: Cmax of metabolite, HAS719 | Predose and 1, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 168, and 192 hours post dose
  Cmax is defined as the maximum observed concentration of drug
PK Parameter: AUC0-t of metabolite, HAS719 | Predose and 1, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 168, and 192 hours post dose
  AUC0-t is defined as the area under the concentration versus time curve from time zero to the last quantifiable concentration
PK Parameter: AUCinf of metabolite, HAS719 | Predose and 1, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 168, and 192 hours post dose
  AUCinf is defined as the area under the concentration versus time curve extrapolated to infinite time

SECONDARY OUTCOMES:
Number of Participants with Adverse Event | up to 38 Days
  Safety will be monitored by vital signs, electrocardiography, and clinical laboratory results
PK Parameter of EQ143: Time to peak concentration (tmax) | Predose and 1, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 168, and 192 hours post dose
PK Parameter of EQ143: elimination half-life (t1/2z) | Predose and 1, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 168, and 192 hours post dose
PK Parameter of EQ143: apparent volume of distribution (Vz/F) | Predose and 1, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 168, and 192 hours post dose
PK Parameter of EQ143: fraction unbound (fu) | Predose and 1, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 168, and 192 hours post dose
PK Parameter of EQ143: unbound peak concentration (Cmaxu) | Predose and 1, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 168, and 192 hours post dose
PK Parameter of EQ143: unbound AUC0-t (AUC0-t U) | Predose and 1, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 168, and 192 hours post dose
PK Parameter of EQ143: unbound apparent clearance (CLu/F) | Predose and 1, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 168, and 192 hours post dose
PK Parameter of metabolite, HAS719: Time to peak concentration (tmax) | Predose and 1, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 168, and 192 hours post dose
PK Parameter of metabolite, HAS719: elimination half-life (t1/2z) | Predose and 1, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 168, and 192 hours post dose
PK Parameter of metabolite, HAS719: apparent volume of distribution (Vz/F) | Predose and 1, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 168, and 192 hours post dose
PK Parameter of metabolite, HAS719: fraction unbound (fu) | Predose and 1, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 168, and 192 hours post dose
PK Parameter of metabolite, HAS719: unbound peak concentration (Cmaxu) | Predose and 1, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 168, and 192 hours post dose
PK Parameter of metabolite, HAS719: unbound AUC0-t (AUC0-t U) | Predose and 1, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 168, and 192 hours post dose
PK Parameter of metabolite, HAS719: unbound apparent clearance (CLu/F) | Predose and 1, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 168, and 192 hours post dose

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - American Institute Research, Los Angeles, California
  - Global Clinical Professionals, St. Petersburg, Florida
  - Texas Liver Institute, San Antonio, Texas